CLINICAL TRIAL: NCT02966431
Title: Effects of a Weight Loss Intervention in College-age Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Strict study protocol and lack of participant reimbursement was not advantageous and feasible as evidenced by the high rate of attrition.
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Jada Stevenson, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT2016JS2
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Experimental): Receive counseling for 8-wks
  Interventions: Behavioral: Counseling
- Control (Placebo Comparator): Does not receive counseling for 8-wks
  Interventions: Behavioral: No Counseling

INTERVENTIONS:
Behavioral: Counseling
  Arms: Counseling
Behavioral: No Counseling
  Arms: Control

SUMMARY:
Determine the effects of an 8-week weight loss intervention.

DETAILED DESCRIPTION:
The purpose of this study is three-fold: 1) Determine whether an 8-week, patient-centered, weight loss intervention can be successfully implemented in overweight, college-age females for promotion of weight loss and prevention of weight regain at 8-weeks, three months, and six months follow-up; 2) Determine the effects of the intervention on established markers of calorie restriction, energy expenditure and body composition; 3) Determine the effects of a liquid meal on physiological and subjective markers of hunger and satiety from pre- to post- 8wk intervention in the intervention group vs control group.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-25years
* Body Mass Index 25.0 to 29.9 kg/m2 (overweight)
* Agree to receive frequent contacts from investigators and communicate with program staff for up to 6 months
* Willing to measure blood glucose via finger prick test three to eight times per day for two weeks
* Able to give written informed consent
* Able to comply with study procedures

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Travel plans that do not permit participation
* Pregnant or planning on becoming pregnant during the 6 months of participation in the study
* Weight loss or gain exceeding 5% of body weight in the past 3 months
* Current participation in a weight loss program
* Diagnosis of mental disorder or chronic disease
* History of eating disorder such as anorexia nervosa, bulimia nervosa, or binge eating disorder (unless approved by program staff)
* History of surgery or procedure that could affect swallowing or digestion
* Any person who is on a medically prescribed diet
* Any current supplement use other than a daily multivitamin
* Any current metabolic medication use other than birth control
* Any bleeding disorders or blood clotting problems
* Anyone who has donated blood or plasma in the last 20 days
* Any tobacco or illicit drug users
* Anyone who has allergies to any of the components of the liquid meal

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Body weight | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No